CLINICAL TRIAL: NCT00350441
Title: A Randomised, Double-Blind, Placebo-Controlled, Single-Centre Study of the Pre-Operative Effect of Sildenafil Citrate on Pulmonary Related Complications Following Cardiopulmonary Bypass in Children Undergoing Cardiac Surgical Repair.
Brief Title: Does Sildenafil Protect Against Pulmonary Related Complications Following Cardiopulmonary Bypass?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow Yorkhill Division (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05/CA/01
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-07

CONDITIONS: Cardiopulmonary Bypass
Keywords: Sildenafil Citrate; Cardiopulmonary bypass; Open heart surgery
MeSH Terms: interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate

SUMMARY:
Does pre-operative administration of Sildenafil (Viagra, Pfizer) reduce the lung injury associated with cardiopulmonary bypass in children undergoing corrective surgical repair of congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

Paediatric patients undergoing open heart surgery utilising cardiopulmonary bypass to correct acyanotic congenital heart disease.

Age > 3 months Parents that show a good understanding of their child's condition and are happy for their child to participate in the study.

Exclusion Criteria:

Patients with known organ dysfunction prior to surgery (pulmonary, renal or hepatic) Communication barrier resulting in poor basic comprehension of the proposed study (e.g. language barrier) Patients with cyanotic heart disease Patients undergoing heart surgery without the use of cardiopulmonary bypass Patients who do not tolerate oral Sildenafil (e.g. Vomiting) or whose surgery is subsequently cancelled.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Tony Vassalos, MB Ch B, Principal Investigator — Royal Hospital for Sick Children
Locations (1):
- Royal Hospital for Sick Children, Glasgow, Strathclyde, United Kingdom